CLINICAL TRIAL: NCT00817258
Title: Phase Ⅱ Study of Concurrent Chemotherapy and Radiotherapy for Stage II Nasopharyngeal Carcinoma
Brief Title: Study of Concurrent Chemotherapy and Radiotherapy for Stage II Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Department of Radiation Oncology,Cancer Hospital, Fudan University, Shanghai, China, Cancer Hospital, Fudan University, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-0701
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Phase 2 Clinical Trial; NPC; radiation therapy; chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): All patients will receive radical radiotherapy with 3D-CRT or IMRT, and cisplatin (40mg/m2) weekly during external radiotherapy.
  Interventions: Drug: cisplatin; Radiation: 3D-CRT (three-dimensional conformal radiation therapy) or IMRT (intensity-modulated radiation therapy)

INTERVENTIONS:
Drug: cisplatin — Cisplatin 40mg/m2,weekly
Radiation: 3D-CRT (three-dimensional conformal radiation therapy) or IMRT (intensity-modulated radiation therapy) — 3D-CRT or IMRT

SUMMARY:
The primary objective of this study is to determine the overall survival in patients with stage II (T1-2N1M0) NPC treated with concurrent chemotherapy and radiotherapy.

Secondary objectives of the study are to evaluate the disease free survival, and distant metastases free survival of patients with stage II NPC treated with this regimen

DETAILED DESCRIPTION:
Radiotherapy alone is the standard treatment for early stage NPC. In retrospective study of early stage NPC patients treated with radiotherapy alone. Patients who had Stage II disease had a worse outcome compared with patients with stage I disease. Chemotherapy, delivered concurrently with radiation therapy, has been adopted as standard treatment for locally advanced NPC. However, concurrent chemoradiation for stage II NPC patients has never been prospectively studied. In the present trial, we hope to assess the value of concurrent chemotherapy and radiotherapy in patients with stage II (T1-2N1) NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven differentiated non-keratinizing carcinoma, and undifferentiated carcinoma of the nasopharynx.
* Stage II disease (T1-2; N1; M0)
* KPS >70
* Age between 18-70
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of > 2000 cells/mm3, platelet count of > 100,000 cells/mm3 (pre treatment without intervention). Bilirubin < 1.5 mg/dl, AST or ALT<2 x upper normal, serum creatinine<1.5mg/dl, creatinine clearance >50ml/min.
* No prior radiation treatment to the head and neck or any prior chemotherapy
* Patients with no prior malignancy (not include basal cell carcinoma of skin)

Exclusion Criteria:

* Evidence of metastases (below the clavicle or distant) by clinical or radiographic examinations.
* Prior radiotherapy to the head and neck region for any reason.
* Initial surgical treatment excluding diagnostic biopsy of the primary site or neck disease.
* Patients with previous or simultaneous primaries, excluding basal cell carcinoma or squamous cell carcinoma of skin.
* Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 and 5 years

SECONDARY OUTCOMES:
disease-free survival, and distant metastases free survival | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Kong, MD, Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University; Chaosu Hu, MD, Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Fudan University, Shanghai, China